CLINICAL TRIAL: NCT04002518
Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the Biomet Cannulated Bone Screw System (Implants and Instrumentation) - A Retrospective/Prospective Study
Brief Title: MDR - Biomet Cannulated Screws
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-35T
Record Dates: First submitted 2019-06-18; First posted 2019-06-28 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Fractures, Bone; Fracture Multiple
MeSH Terms: conditions — Fractures, Bone; Fractures, Multiple

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Small Screws: Patients who have surgically been treated with a 3.0mm or 4.0mm screw.
  Interventions: Device: Biomet Cannulated Screw: 3.0, 4.0, 5.0, 6.5, and 8.0mm screws.
- Large Screws: Patients who have surgically been treated with a 5.0mm, 6.5mm or 8.0mm screw.
  Interventions: Device: Biomet Cannulated Screw: 3.0, 4.0, 5.0, 6.5, and 8.0mm screws.

INTERVENTIONS:
Device: Biomet Cannulated Screw: 3.0, 4.0, 5.0, 6.5, and 8.0mm screws. — Treatment of identified conditions, i.e. fracture fixation, arthrodesis, osteotomy, with a cannulated screw.

SUMMARY:
The objective of this retrospective enrollment/prospective follow up study is to collect data confirming safety, performance, and clinical benefits of the Biomet Cannulated Bone Screw System (Implants and Instrumentation) when used according to the approved Indications for Use (IFU).

DETAILED DESCRIPTION:
The objective of this retrospective enrollment/prospective follow up study is to collect data confirming safety, performance, and clinical benefits of the Biomet Cannulated Bone Screw System (Implants and Instrumentation) when used according to the approved Indications for Use (IFU).

Safety will be established by recording the incidence and frequency of complications and adverse events. Relationship of the events to either implant or instrumentation should be specified.

Performance and clinical benefits will be assessed by analyzing fracture healing/fusion and the overall pain and functional performance of subjects who received the Biomet Cannulated Bone Screws by recording survey questions. Zimmer Biomet defines the expected performance rate for Cannulated Screws for long and small bone fractures to be a union rate of at least 81% at 8-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older.

All patients operated on for the following indications:

* Group 1, Small Cannulated Screws (4.0mm and smaller diameter) are intended for use in:

  1. Fixation of small bones, including those in the foot, patella, ankle, wrist and elbow.
  2. Arthrodesis of the foot, wrist and elbow.
  3. Small and long bone osteotomies.
  4. Fracture fixation of small bones, small bone fragments and long bones.
* Group 2, Large Cannulated Screws (5mm and larger in diameter) are intended for use in:

  1. Fixation of fractures in long bones and long bone fragments.
  2. Long bone osteotomies (femur, tibia, foot, ankle, olecranon).
  3. Arthrodesis and fracture fixation of the foot and ankle, such as Jones fractures of the fifth metatarsal, and Calcaneal fractures.
* Group 3, Large Cannulated Screws (6.5mm and larger in diameter) are intended for use in:

  1. Slipped capital femoral epiphysis
  2. Pediatric femoral neck fractures
  3. Tibial plateau fractures
  4. SI joint disruptions
  5. Intercondylar femur fractures
  6. Subtalar arthrodesis
  7. Fixation of pelvis and iliosacral joint
* Patients must have the ability and willingness to follow instructions, including control of weight and activity levels.
* Patient must have a good nutritional state.

Exclusion Criteria:

* Infections.
* Patient conditions including blood supply limitations, insufficient quantity or quality of bone.
* Patients with mental or neurologic conditions who are unwilling or incapable fo following postoperative care instructions.
* Foreign body sensitivity where material sensitivity is suspected or unknown, testing is to be completed prior to implantation of the device.
* Patient is a prisoner.
* Patient is a current alcohol or drug abuser.
* Patient is known to be pregnant or breastfeeding.
* Patient has a psychiatric illness or cognitive deficit that will not allow for proper informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study populations will be a consecutive series of subjects that have received the Biomet Cannulated Screw. Patients will be enrolled into one of the two identified groups: Small Screws (3.0mm and 4.0mm), or Large Screws (5.0mm, 6.5mm and 8.0mm).
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Device Safety Assessed Through the Incidence and Frequency of Revisions, Complications, and Adverse Events | Out to12+ months
  Assessment of safety by recording and analyzing the incidence and frequency of revisions, complications, and adverse events.

SECONDARY OUTCOMES:
Device Performance and Clinical Benefits Assessed by a Patient Questionnaire Case Report Form | Out to 12+ months
  Performance and clinical benefits demonstrated by the assessment of survey questions.
Device Performance and Clinical Benefits Assessed by a Follow-Up Analysis Case Report Form | Out to 12+ months
  Performance and clinical benefits demonstrated by the assessment of fracture healing/fusion and survey questions.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (3):
- United States (3):
  - Zimmer Biomet, Warsaw, Indiana
  - Orthopedic Foot and Ankle Center, Worthington, Ohio
  - Associated Foot & Ankle Centers of Northern Virginia, Lake Ridge, Virginia

IPD SHARING:
Plan to Share IPD: No